CLINICAL TRIAL: NCT04358263
Title: Comparison of CGM in Randomised Study of Real-time and Intermittently-scanned Systems in T1D With Normal Awareness of Hypoglycemia (CORRIDA)
Brief Title: Is Real-time CGM Superior to Flash Glucose Monitoring
Acronym: CORRIDA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jan Soupal, MD, Principal Investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CORRIDA
Record Dates: First submitted 2020-04-15; First posted 2020-04-24 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Continuous Glucose Monitoring; Flash Glucose Monitoring; Hypoglycemia; Time in Range; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- rtCGM (Experimental): Patients with use of the Guardian Connect Mobile system (real-time continuous glucose monitoring).
  Interventions: Device: Continuous Glucose Monitoring Guardian Connect Mobile system (real-time continuous glucose monitoring)
- isCGM (Experimental): Patients with use of the FreeStyle Libre Flash system (intermittently-scanned continuous glucose monitoring).
  Interventions: Device: Continuous Glucose Monitoring FreeStyle Libre Flash system (intermittently-scanned continuous glucose monitoring)

INTERVENTIONS:
Device: Continuous Glucose Monitoring Guardian Connect Mobile system (real-time continuous glucose monitoring) — rtCGM and isCGM are used in Type 1 diabetic patients to improve glucose control and to minimize or avoid severe hypoglycaemia.
  Arms: rtCGM
Device: Continuous Glucose Monitoring FreeStyle Libre Flash system (intermittently-scanned continuous glucose monitoring) — rtCGM and isCGM are used in Type 1 diabetic patients to improve glucose control and to minimize or avoid severe hypoglycaemia.
  Arms: isCGM

SUMMARY:
The aim of the investigator's study is to compare real-time continuous glucose monitoring and flash glucose monitoring in adult patients with Type 1 Diabetes during 4-day training program focused on physical activity and over 4 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients with T1D naive to rtCGM and isCGM
* Type 1 diabetes for >2 years
* ≥ 18 years old
* CSII or MDI
* GOLD score < 4, no history of severe hypoglycemia within last 6 month
* written informed consent prior to starting study related activity

Exclusion Criteria:

* severe noncompliance
* severe diabetic retinopathy and/or macular edema
* lactation, pregnancy, intending to become pregnant during study
* condition likely to require MRI
* use of acetaminophen-containing medication
* unwillingness to use the study device for >70% of time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of time in hypoglycemic ranges | Up to 2 months
  <3,9 mmol/L (70 mg/dl) and <3,0 mmol/L (54 mg/dl)

SECONDARY OUTCOMES:
Percentage of time in target ranges | Up to 2 months
  3,9-10,0 mmol/L (70-180 mg/dl)
Percentage of time in hyperglycemic ranges | Up to 2 months
  (>10,0 mmol/L (180 mg/dl) and >13,9 mmol/L (250 mg/dl)
Changes in glycemic variability | Up to 2 months
  Expressed as the coefficient of variation
Mean sensor glucose concentration | Up to 2 months
  Measured by rtCGM or isCGM
Changes in quality of life as assessed by validated questionnaire | Up to 2 months
  Assessed by The World Health Organization Quality of Life (WHOQOL)-BREF (Field Trial Version).
  This questionnaire contains in total 26 questions in four Domains (Physical health, Psychological health, Social relationships, Environment). Scores in total range between 4-20 (each Domain 0-5), higher scores denote higher quality of life.
Incidence of severe hypoglycaemia | Up to 2 months
  Requiring third-party assistance to treat
Changes in glycated haemoglobin (HbA1c) | Up to 2 months
  Differences between HbA1c values in the initial period and after follow-up and differences of HbA1c between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Soupal, Principal Investigator — Charles University, Prague
Locations (1):
- 3rd Department of Internal Medicine, 1st Faculty of Medicine Charles University, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cryer PE. Hypoglycemia: still the limiting factor in the glycemic management of diabetes. Endocr Pract. 2008 Sep;14(6):750-6. doi: 10.4158/EP.14.6.750. PMID 18996798
- [Background] Moser O, Tschakert G, Mueller A, Groeschl W, Pieber TR, Obermayer-Pietsch B, Koehler G, Hofmann P. Effects of High-Intensity Interval Exercise versus Moderate Continuous Exercise on Glucose Homeostasis and Hormone Response in Patients with Type 1 Diabetes Mellitus Using Novel Ultra-Long-Acting Insulin. PLoS One. 2015 Aug 28;10(8):e0136489. doi: 10.1371/journal.pone.0136489. eCollection 2015. PMID 26317981
- [Background] Cryer PE. Hypoglycemia in type 1 diabetes mellitus. Endocrinol Metab Clin North Am. 2010 Sep;39(3):641-54. doi: 10.1016/j.ecl.2010.05.003. PMID 20723825
- [Background] Edelman SV, Argento NB, Pettus J, Hirsch IB. Clinical Implications of Real-time and Intermittently Scanned Continuous Glucose Monitoring. Diabetes Care. 2018 Nov;41(11):2265-2274. doi: 10.2337/dc18-1150. PMID 30348844
- [Background] Beck RW, Riddlesworth T, Ruedy K, Ahmann A, Bergenstal R, Haller S, Kollman C, Kruger D, McGill JB, Polonsky W, Toschi E, Wolpert H, Price D; DIAMOND Study Group. Effect of Continuous Glucose Monitoring on Glycemic Control in Adults With Type 1 Diabetes Using Insulin Injections: The DIAMOND Randomized Clinical Trial. JAMA. 2017 Jan 24;317(4):371-378. doi: 10.1001/jama.2016.19975. PMID 28118453
- [Background] Soupal J, Petruzelkova L, Flekac M, Pelcl T, Matoulek M, Dankova M, Skrha J, Svacina S, Prazny M. Comparison of Different Treatment Modalities for Type 1 Diabetes, Including Sensor-Augmented Insulin Regimens, in 52 Weeks of Follow-Up: A COMISAIR Study. Diabetes Technol Ther. 2016 Sep;18(9):532-8. doi: 10.1089/dia.2016.0171. Epub 2016 Aug 2. PMID 27482825
- [Background] Soupal J, Petruzelkova L, Grunberger G, Haskova A, Flekac M, Matoulek M, Mikes O, Pelcl T, Skrha J Jr, Horova E, Skrha J, Parkin CG, Svacina S, Prazny M. Glycemic Outcomes in Adults With T1D Are Impacted More by Continuous Glucose Monitoring Than by Insulin Delivery Method: 3 Years of Follow-Up From the COMISAIR Study. Diabetes Care. 2020 Jan;43(1):37-43. doi: 10.2337/dc19-0888. Epub 2019 Sep 17. PMID 31530663
- [Background] Oskarsson P, Antuna R, Geelhoed-Duijvestijn P, Krӧger J, Weitgasser R, Bolinder J. Impact of flash glucose monitoring on hypoglycaemia in adults with type 1 diabetes managed with multiple daily injection therapy: a pre-specified subgroup analysis of the IMPACT randomised controlled trial. Diabetologia. 2018 Mar;61(3):539-550. doi: 10.1007/s00125-017-4527-5. Epub 2017 Dec 23. PMID 29273897
- [Background] Reddy M, Jugnee N, Anantharaja S, Oliver N. Switching from Flash Glucose Monitoring to Continuous Glucose Monitoring on Hypoglycemia in Adults with Type 1 Diabetes at High Hypoglycemia Risk: The Extension Phase of the I HART CGM Study. Diabetes Technol Ther. 2018 Nov;20(11):751-757. doi: 10.1089/dia.2018.0252. Epub 2018 Sep 28. PMID 30265562
- [Derived] Haskova A, Radovnicka L, Petruzelkova L, Parkin CG, Grunberger G, Horova E, Navratilova V, Kade O, Matoulek M, Prazny M, Soupal J. Real-time CGM Is Superior to Flash Glucose Monitoring for Glucose Control in Type 1 Diabetes: The CORRIDA Randomized Controlled Trial. Diabetes Care. 2020 Nov;43(11):2744-2750. doi: 10.2337/dc20-0112. Epub 2020 Aug 28. PMID 32859607